CLINICAL TRIAL: NCT05994729
Title: Impact of Renal Denervation in Patients With Coronary Microvascular Dysfunction: Study Design and Rationale
Acronym: IMPRESSION
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Aurelia Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AH Card. 08-23
Record Dates: First submitted 2023-08-09; First posted 2023-08-16 (Actual); Last update posted 2023-10-24 (Actual); Status verified 2023-10

CONDITIONS: Coronary Microvascular Dysfunction; Resistant Hypertension; Hypertensive Heart Disease
Keywords: MVD; HHD

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Candidates to RDN with ascertained CMD (Experimental): Patients that are candidates to receive RDN for resistant/difficult to control hypertension, who also have documented coronary microvascular dysfunction
  Interventions: Diagnostic Test: Invasive Physiological Assessment of Coronary Circulation

INTERVENTIONS:
Diagnostic Test: Invasive Physiological Assessment of Coronary Circulation — After 2 months long rule-in phase required to exclude the unsuitable patients, study population will undergo RDN as indicated to treat resistant or difficult to control hypertension; 12 months after RDN, they will undergo invasive physiological study, comprehensive of Coronary Flow Reserve, Index of Microvascular Resistance, Mean Transit Time. These data will be then compared to the baseline ones obtained during the screening phase.
  Other Names: CFR; IMR; Tmn

SUMMARY:
Long-standing hypertension may cause an impairment in microvascular coronary circulation which is involved in many different cardiac conditions. Renal denervation (RDN) has been successfully proven as a valuable and powerful therapeutic choice to consider for patients with resistant hypertension; moreover this procedure looks promising in other cardiac disease such as heart failure and atrial fibrillation, given its ability to downregulate sympathetic nervous system The aim of this study is to explore the effect of renal denervation and blood pressure control on coronary microvascular dysfunction.

This is a multicenter, prospective, non randomized, open-label, interventional study. Consecutive patients with resistant hypertension, non obstructive coronary artery disease and documented microvascular dysfunction will be enrolled. Patients will undergo renal denervation by Spyral Symplicity 3 and re-assessment of coronary microvascular function 12 months after the procedure. Primary endpoint will be the difference in average index of microcirculatory resistance value.

DETAILED DESCRIPTION:
The aim of this study is to evaluate the effect of radiofrequency RDN performed with Spyral Symplicity 3 on microvascular function in patients with ascertained hypertension related coronary microvascular dysfunction (hy-CMD) and/or hypertensive cardiomyopathy. Our hypothesis is that RDN could improve invasive parameters of microvascular function in patients with hy-CMD; these would mean that RDN would be able to at least partially revert the pathogenesis of hy-CMD.

The study design comprises an initial rule-in and enrollment phase, required to properly select the target population, followed by the actual study procedural phase.

Patients amenable to RDN will be hospitalized and enter the rule-in phase to check for eligibility.

Before performing the actual RDN, patients will be asked for the written informed consent to receive physiological evaluation.

Only patients that will be diagnosed with hy-CMD will eventually enter the actual study phase.

This phase will comprise repeated outpatients visits, according to a predetermined schedule, including a new hospitalization at 12 months to reassess coronary microvascular physiology.

ELIGIBILITY:
Rul-in Phase Inclusion Criteria:

* Non obstructive stable coronary artery disease (CAD) on invasive coronary angiography (defined as the absence of either >50% angiographic stenosis or any flow limiting lesion on functional evaluation)
* Suspected diagnosis of difficult to control/ resistant hypertension for which renal denervation by radiofrequency ablation with Spyral Symplicity 3 could be considered.

Rule-in Phase Exclusion Criteria:

* Initiation of either nitrates, beta-blocker or calcium channel blocker less than 30 days before the end of the rule-in phase
* Physiological assessment performed during first medical contact documenting preserved coronary microvascular function
* Physiological assessment performed at the "first contact" hospitalization followed by modification of medical therapy during the rule-in phase, before RDN
* Acceptable blood pressure control after medical treatment optimization
* Identification of secondary causes of hypertension
* Renal artery anatomy not suitable for RDN
* Ejection fraction below 30%
* Life expectancy below 1 year
* Indication to cardiac surgery
* Adenosine allergy
* Pregnancy
* Large necrotic area documented by either MRI, SPECT or combination of ECG signs + Echocardiographic images.
* Hemodynamic instability
* Refuse to sign informed consent
* Age below 18 or above 80

Study Phase Inclusion Criteria:

* Having coronary microvascular dysfunction documented by invasive functional assessment (IMR>25 and or CFR < 2)
* Fulfilling all the rule-in phase inclusion criteria without any rule-in phase exclusion criteria

Study Phase Exclusion Criteria:

* Refuse to sign informed consent
* Evidence of newly detected obstructive CAD on invasive coronary angiography performed 6 months after RDN

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 87 (Estimated)
Dates: Start 2024-01-01 (Estimated); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Index of microvascular resistance (IMR) | 12 months
  Matched comparison of IMR from baseline to 12 months after RDN

SECONDARY OUTCOMES:
Coronary Flow Reserve (CFR) | 12 months
  Matched comparison of CFR from baseline to 12 months after RDN
Mean transit time (TMN) | 12 months
  Matched comparison of both resting and hyperemic TMN from baseline to 12 months after RDN
Systolic Blood Pressure (BP) on Ambulatory blood pressure monitoring (ABPM) | 12 Months
  Matched Comparison of Average Systolic Blood Pressure measured on 24 hour Ambulatory Blood Pressure Monitoring
Diastolic BP on ABPM | 12 Months
  Matched Comparison of Average Systolic Blood Pressure measured on 24 hour Ambulatory Blood Pressure Monitoring
Average BP on ABPM | 12 Months
  Matched Comparison of Average Mean Blood Pressure measured on 24 hour Ambulatory Blood Pressure Monitoring
Time in Therapeutic BP Range | 12 Months
  Matched Comparison of total time spent with both systolic and diastolic BP within normality range measured on 24 hour Ambulatory Blood Pressure Monitoring
BP Medication Burden | 12 Months
  Matched Comparison of Total Number of BP medication prescribed to the subject
Mini-SAQ Score (Seattle Angina Questionnaire) | 12 Months
  Matched Comparison of Average Score on Mini Seattle Angina Questionnaire (SAQ)
NTproBNP | 12 Months
  Matched Comparison of Average NTproBNP

CONTACTS AND LOCATIONS:
Overall Officials: Fabrizio Tomai, MD, FACC, FESC, Principal Investigator — Aurelia Hospital; stefano migliaro, MD, Study Chair — Aurelia Hospital